CLINICAL TRIAL: NCT01453712
Title: Prospective Randomized Trial On Radiation Dose Estimates Of CT Angiography In Patients Applying Iterative Image Reconstruction Techniques - The PROTECTION V Study -
Acronym: PROTECTION-V
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE-DHM-PROTV
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary CT angiography; radiation dose; iterative image reconstruction; detection
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Conventional coronary CT angiography using standard reconstruction technique (filtered back projection).
  Interventions: Radiation: Control group
- Intervention group (Experimental): Using the new scan protocol with 30 % less tube current and iterative image reconstruction algorithm.
  Interventions: Radiation: Intervention group

INTERVENTIONS:
Radiation: Control group — Conventional coronary CT angiography using standard reconstruction technique (filtered back projection).
  Arms: Control group
Radiation: Intervention group — Using the new scan protocol with 30 % less tube current and iterative image reconstruction algorithm.
  Arms: Intervention group

SUMMARY:
The objective of this study is to compare a standard coronary CT angiography scan protocol with conventional image reconstruction with a scan protocol using reduced tube current and a new image reconstruction algorithm. The investigators hypothesize that the image quality of the new scan protocol is not inferior, while radiation dose estimates are reduced by around 30%.

Secondary endpoints of the study include quantitative image quality parameters, prevalence of non-diagnostic studies, prevalence of coronary artery plaques and plaque characteristics (calcified, non-calcified, mixed) and prevalence of follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

1. patients with an indication for a coronary CT angiography (planned evaluation of the coronary arteries)
2. signed informed consent
3. stable sinus rhythm
4. age > 18 years

Exclusion Criteria:

1. known allergy to contrast agents.
2. patients with known coronary artery disease
3. pregnancy
4. no stable sinus rhythm
5. coronary ct examinations not focussing on coronary arteries

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Image quality | 1 month
  Compared with a conventional scan protocol the use of a new scan protocol using iterative image reconstruction and reduced tube current is associated with a comparable diagnostic image quality, while the radiation dose estimates are significantly reduced.

SECONDARY OUTCOMES:
Quantitative image quality parameters | 1 month
  Quantitative image quality parameters, e.g. image noise, signal and contrast intensity, signal- and contrast-to-noise-ratios
Prevalence of non-diagnostic examinations | 1 month
  Prevalence of non-diagnostic examinations in both study arms.
Prevalence of coronary artery plaques | 1 month
  Prevalence of coronary artery plaques and coronary artery plaques characteristics (non-calcified, calcified, mixed) in both study arms.
Prevalence of follow-up examinations | 1 month
  Prevalence of follow-up examinations in both study arms.
Radiation dose | 1 month
  Radiation dose in both study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Deseive S, Chen MY, Korosoglou G, Leipsic J, Martuscelli E, Carrascosa P, Mirsadraee S, White C, Hadamitzky M, Martinoff S, Menges AL, Bischoff B, Massberg S, Hausleiter J. Prospective Randomized Trial on Radiation Dose Estimates of CT Angiography Applying Iterative Image Reconstruction: The PROTECTION V Study. JACC Cardiovasc Imaging. 2015 Aug;8(8):888-96. doi: 10.1016/j.jcmg.2015.02.024. Epub 2015 Jul 15. PMID 26189118